CLINICAL TRIAL: NCT01709578
Title: A Randomized, Double-blind, Parallel, Placebo-controlled Study Assessing the Efficacy and Safety of Sarilumab Added to Non-biologic DMARD Therapy in Patients With Rheumatoid Arthritis Who Are Inadequate Responders to or Intolerant of TNF-α Antagonists
Brief Title: To Evaluate The Effect Of SAR153191 (REGN88) Added To Other RA Drugs In Patients With RA Who Are Not Responding To Or Intolerant Of Anti-TNF Therapy (SARIL-RA-TARGET)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC10832; U1111-1115-8466 (Other: UTN); 2011-003538-16 (EudraCT Number)
Record Dates: First submitted 2012-10-15; First posted 2012-10-18 (Estimated); Results first posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab; Hydroxychloroquine; Methotrexate; Sulfasalazine; Leflunomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo q2w (Placebo Comparator): Placebo matched to sarilumab once every 2 weeks (q2w) was added to one or a combination of the nonbiologic DMARD (hydroxychloroquine, methotrexate, sulfasalazine and/or Leflunomide), except for simultaneous combination use of leflunomide and methotrexate for 24 weeks.
  Interventions: Drug: placebo; Drug: hydroxychloroquine; Drug: methotrexate; Drug: sulfasalazine; Drug: leflunomide
- Sarilumab 150 mg q2w (Experimental): Sarilumab 150 mg q2w was added to one or a combination of the nonbiologic DMARD (hydroxychloroquine, methotrexate, sulfasalazine and/or Leflunomide), except for simultaneous combination use of leflunomide and methotrexate for 24 weeks.
  Interventions: Drug: Sarilumab; Drug: hydroxychloroquine; Drug: methotrexate; Drug: sulfasalazine; Drug: leflunomide
- Sarilumab 200 mg q2w (Experimental): Sarilumab 200 mg q2w was added to one or a combination of the nonbiologic DMARD (hydroxychloroquine, methotrexate, sulfasalazine and/or Leflunomide), except for simultaneous combination use of leflunomide and methotrexate for 24 weeks.
  Interventions: Drug: Sarilumab; Drug: hydroxychloroquine; Drug: methotrexate; Drug: sulfasalazine; Drug: leflunomide

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form:solution Route of administration: subcutaneous
  Other Names: SAR153191; REGN88
  Arms: Sarilumab 150 mg q2w; Sarilumab 200 mg q2w
Drug: placebo — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Placebo q2w
Drug: hydroxychloroquine — Dispensed according to the local practice.
Drug: methotrexate — Dispensed according to the local practice.
Drug: sulfasalazine — Dispensed according to the local practice.
Drug: leflunomide — Dispensed according to the local practice.

SUMMARY:
Primary Objective:

To demonstrate that sarilumab added to disease modifying anti-rheumatic drugs (DMARDs) were effective for:

* reduction of signs and symptoms at Week 24 and
* improvement of physical function at Week 12

in participants with active rheumatoid arthritis (RA) who were inadequate responders or intolerant to tumor necrosis factor alpha (TNF-α) antagonists.

Secondary Objectives:

The secondary objectives were to investigate the effects of SAR153191 (REGN88) when added to DMARD therapy, in participants with active RA who were inadequate responders or intolerant to TNF-α antagonists, for:

* Reduction of signs and symptoms at Week 12;
* Improvement in physical function at Week 24;
* Improvement in disease activity score as measured by other American College of Rheumatology (ACR) derived components at Weeks 12 and 24;
* Improvement in quality of life as measured by participant reported outcomes (PROs) at intermediate visits and Week 24.

To assess the exposure of sarilumab added to DMARD therapy in this population.

To assess the safety of sarilumab in this population.

DETAILED DESCRIPTION:
Total study duration was up to 34 weeks: screening up to 28 days, treatment phase of 24 weeks, and post-treatment follow-up of 6 weeks.

After completion of the treatment phase of this study, participant were eligible to enter a long term safety study (LTS11210) for active treatment with SAR153191 (REGN88).

ELIGIBILITY:
Inclusion criteria:

Diagnosis of RA ≥6 months duration, according to the ACR /European League against Rheumatism (EULAR) 2010 RA Classification Criteria

ACR Class I-III functional status, based on 1991 revised criteria

Anti-TNF therapy failures, defined by the investigator as participants with an inadequate clinical response, after being treated for at least 3 consecutive months, and/or intolerance to at least 1 anti-TNF blocker(s), resulting in or requiring their discontinuation:

* TNF-blockers included, but were not limited to, etanercept, infliximab, adalimumab, golimumab and/or certolizumab

Moderate-to-severely active RA

Continuous treatment with one or a combination of DMARDs (except for simultaneous combination use of leflunomide and methotrexate) for at least 12 weeks prior to baseline and on a stable dose(s) for at least 6 weeks prior to screening:

* Methotrexate - 6 to 25 mg/week orally or parenterally
* Leflunomide - 10 to 20 mg orally daily
* Sulfasalazine - 1000 to 3000 mg orally daily
* Hydroxychloroquine - 200 to 400 mg orally daily

Exclusion criteria:

Participants <18 years of age or legal adult age

Past history of, or current, autoimmune or inflammatory systemic or localized joint disease(s) other than RA

History of juvenile idiopathic arthritis or arthritis onset prior to age 16

Severe active systemic RA, including but not limited to vasculitis, pulmonary fibrosis, and/or Felty's syndrome.

Treatment with anti-TNF agents, as follows:

* Within 28 days prior to the baseline visit - etanercept
* Within 42 days prior to the baseline visit - infliximab, adalimumab, golimumab, certolizumab pegol

Treatment with previous RA-directed biologic agents with other than TNF antagonist mechanisms:

Within 28 days prior to the randomization (baseline) visit - anakinra Within 42 days prior to the randomization (baseline) visit - abatacept

Within 6 months prior to the randomization (baseline) visit - any cell depleting agents including but not limited to rituximab without a normal lymphocyte and cluster of differentiation (CD) 19+ lymphocyte count

Treatment with any DMARD other than those allowed per protocol and limited to the maximum specified dosage within 12 weeks prior to baseline

Treatment with prednisone >10 mg or equivalent per day, or change in dosage within 4 weeks prior to baseline visit

Any parenteral or intra-articular glucocorticoid injection within 4 weeks prior to baseline

Prior treatment with anti-interleukin (IL) -6 or IL-6 receptor antagonist therapies, including tocilizumab or sarilumab, participation in a prior study of sarilumab, irrespective of treatment arm

Prior treatment with a Janus kinase inhibitor (such as tofacitinib)

New treatment or dose-adjustment to ongoing medication for dyslipidemia within 6 weeks prior to randomization, ie, stable dose for at least 6 weeks prior to randomization

Participation in any clinical research study evaluating another investigational drug or therapy within 5 half-lives or 60 days of first investigational medicinal product (IMP) administration, whichever was longer

History of alcohol or drug abuse within 5 years prior to the screening visit

Participants with a history of malignancy other than adequately-treated carcinoma in-situ of the cervix, nonmetastatic squamous cell or basal cell carcinoma of the skin, within 5 years prior to the randomization (baseline) visit. Nonmalignant lymphoproliferative disorders were also excluded

Participants with active tuberculosis or latent tuberculosis infection

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (196):
- United States (56):
  - Investigational Site Number 840070, Anniston, Alabama
  - Investigational Site Number 840138, Birmingham, Alabama
  - Investigational Site Number 840142, Phoenix, Arizona
  - Investigational Site Number 840134, Fullerton, California
  - Investigational Site Number 840141, Glendale, California
  - Investigational Site Number 840111, La Jolla, California
  - Investigational Site Number 840135, San Diego, California
  - Investigational Site Number 840021, Santa Maria, California
  - Investigational Site Number 840100, Stanford, California
  - Investigational Site Number 840049, Upland, California
  - Investigational Site Number 840131, Whittier, California
  - Investigational Site Number 840201, Denver, Colorado
  - Investigational Site Number 840130, Lewes, Delaware
  - Investigational Site Number 840125, DeBary, Florida
  - Investigational Site Number 840048, Miami, Florida
  - Investigational Site Number 840024, Naples, Florida
  - Investigational Site Number 840006, Orlando, Florida
  - Investigational Site Number 840128, Ormond Beach, Florida
  - Investigational Site Number 840063, Palm Harbor, Florida
  - Investigational Site Number 840060, Sarasota, Florida
  - Investigational Site Number 840140, Tampa, Florida
  - Investigational Site Number 840126, Vero Beach, Florida
  - Investigational Site Number 840018, Idaho Falls, Idaho
  - Investigational Site Number 840110, Meridian, Idaho
  - Investigational Site Number 840052, Kansas City, Kansas
  - Investigational Site Number 840015, Lexington, Kentucky
  - Investigational Site Number 840120, Baton Rouge, Louisiana
  - Investigational Site Number 840109, Lake Charles, Louisiana
  - Investigational Site Number 840055, Frederick, Maryland
  - Investigational Site Number 840150, Lansing, Michigan
  - Investigational Site Number 840137, Saint Clair Shores, Michigan
  - Investigational Site Number 840037, Tupelo, Mississippi
  - Investigational Site Number 840112, Lincoln, Nebraska
  - Investigational Site Number 840106, Orchard Park, New York
  - Investigational Site Number 840121, Rochester, New York
  - Investigational Site Number 840115, Roslyn, New York
  - Investigational Site Number 840118, Smithtown, New York
  - Investigational Site Number 840139, Syracuse, New York
  - Investigational Site Number 840123, Charlotte, North Carolina
  - Investigational Site Number 840116, Wilmington, North Carolina
  - Investigational Site Number 840127, Oklahoma City, Oklahoma
  - Investigational Site Number 840011, Tulsa, Oklahoma
  - Investigational Site Number 840009, Duncansville, Pennsylvania
  - Investigational Site Number 840117, Pittsburgh, Pennsylvania
  - Investigational Site Number 840062, Reading, Pennsylvania
  - Investigational Site Number 840058, Columbia, South Carolina
  - Investigational Site Number 840025, Jackson, Tennessee
  - Investigational Site Number 840059, Memphis, Tennessee
  - Investigational Site Number 840132, Austin, Texas
  - Investigational Site Number 840022, Dallas, Texas
  - Investigational Site Number 840114, El Paso, Texas
  - Investigational Site Number 840133, Houston, Texas
  - Investigational Site Number 840129, Houston, Texas
  - Investigational Site Number 840074, Mesquite, Texas
  - Investigational Site Number 840036, Spokane, Washington
  - Investigational Site Number 840124, Clarksburg, West Virginia
- Argentina (11):
  - Investigational Site Number 032015, Buenos Aires
  - Investigational Site Number 032008, Buenos Aires
  - Investigational Site Number 032019, Caba
  - Investigational Site Number 032006, Caba
  - Investigational Site Number 032016, Capital Federal
  - Investigational Site Number 032020, Córdoba
  - Investigational Site Number 032017, La Plata
  - Investigational Site Number 032010, Ramos Mejía
  - Investigational Site Number 032013, Rosario
  - Investigational Site Number 032004, San Miguel de Tucumán
  - Investigational Site Number 032009, Zárate
- Investigational Site Number 036014, Victoria Park, Australia
- Austria (2):
  - Investigational Site Number 040004, Stockerau
  - Investigational Site Number 040003, Vienna
- Brazil (6):
  - Investigational Site Number 076001, Curitiba
  - Investigational Site Number 076016, Curitiba
  - Investigational Site Number 076006, Goiânia
  - Investigational Site Number 076010, Juiz de Fora
  - Investigational Site Number 076005, Rio de Janeiro
  - Investigational Site Number 076015, Rio de Janeiro
- Canada (3):
  - Investigational Site Number 124005, Toronto
  - Investigational Site Number 124009, Trois-Rivières
  - Investigational Site Number 124104, Victoria
- Investigational Site Number 152015, Temuco, Chile
- Colombia (7):
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170006, Bogotá
  - Investigational Site Number 170012, Bogotá
  - Investigational Site Number 170007, Bucaramanga
  - Investigational Site Number 170009, Bucaramanga
  - Investigational Site Number 170014, Chía
  - Investigational Site Number 170019, Medellín
- Czechia (5):
  - Investigational Site Number 203008, Hostivice
  - Investigational Site Number 203004, Ostrava
  - Investigational Site Number 203007, Prague
  - Investigational Site Number 203002, Uherské Hradiště
  - Investigational Site Number 203006, Zlín
- Ecuador (3):
  - Investigational Site Number 218003, Cuenca
  - Investigational Site Number 218001, Guayaquil
  - Investigational Site Number 218002, Quito
- Germany (13):
  - Investigational Site Number 276011, Bad Nauheim
  - Investigational Site Number 276010, Berlin
  - Investigational Site Number 276001, Berlin
  - Investigational Site Number 276014, Berlin
  - Investigational Site Number 276018, Deggingen
  - Investigational Site Number 276004, Erlangen
  - Investigational Site Number 276015, Halle
  - Investigational Site Number 276013, Hamburg
  - Investigational Site Number 276016, Leipzig
  - Investigational Site Number 276017, München
  - Investigational Site Number 276021, Osnabrück
  - Investigational Site Number 276020, Tübingen
  - Investigational Site Number 276019, Zerbst
- Greece (2):
  - Investigational Site Number 300002, Heraklion
  - Investigational Site Number 300005, Thessaloniki
- Guatemala (3):
  - Investigational Site Number 320002, Guatemala City
  - Investigational Site Number 320003, Guatemala City
  - Investigational Site Number 320001, Guatemala City
- Hungary (4):
  - Investigational Site Number 348022, Budapest
  - Investigational Site Number 348003, Debrecen
  - Investigational Site Number 348004, Veszprém
  - Investigational Site Number 348017, Veszprém
- Israel (3):
  - Investigational Site Number 376001, Haifa
  - Investigational Site Number 376003, Petah Tikva
  - Investigational Site Number 376002, Tel Litwinsky
- Italy (5):
  - Investigational Site Number 380011, Catania
  - Investigational Site Number 380002, Florence
  - Investigational Site Number 380005, Genova
  - Investigational Site Number 380014, Milan
  - Investigational Site Number 380013, Udine
- Lithuania (3):
  - Investigational Site Number 440005, Kaunas
  - Investigational Site Number 440006, Klaipėda
  - Investigational Site Number 440007, Vilnius
- Mexico (10):
  - Investigational Site Number 484023, Chihuahua City
  - Investigational Site Number 484018, Guadalajara
  - Investigational Site Number 484002, Guadalajara
  - Investigational Site Number 484024, Guadalajara
  - Investigational Site Number 484010, Mexicali
  - Investigational Site Number 484017, México
  - Investigational Site Number 484019, Monterrey
  - Investigational Site Number 484020, Monterrey
  - Investigational Site Number 484005, Monterrey
  - Investigational Site Number 484021, Querétaro
- New Zealand (5):
  - Investigational Site Number 554005, Hamilton
  - Investigational Site Number 554011, Nelson
  - Investigational Site Number 554007, Otahuhu
  - Investigational Site Number 554001, Timaru
  - Investigational Site Number 554006, Wellington
- Peru (10):
  - Investigational Site Number 604010, Lima
  - Investigational Site Number 604009, Lima
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604012, Lima
  - Investigational Site Number 604013, Lima
  - Investigational Site Number 604001, Lima
  - Investigational Site Number 604008, Lima
  - Investigational Site Number 604007, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604014, Lima
- Poland (8):
  - Investigational Site Number 616014, Bialystok
  - Investigational Site Number 616019, Bydgoszcz
  - Investigational Site Number 616015, Elblag
  - Investigational Site Number 616018, Poznan
  - Investigational Site Number 616016, Szczecin
  - Investigational Site Number 616004, Warsaw
  - Investigational Site Number 616017, Warsaw
  - Investigational Site Number 616020, Wroclaw
- Portugal (3):
  - Investigational Site Number 620002, Lisbon
  - Investigational Site Number 620004, Lisbon
  - Investigational Site Number 620007, Ponte de Lima
- Romania (4):
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642012, Bucharest
  - Investigational Site Number 642002, Bucharest
  - Investigational Site Number 642014, Iași
- Russia (5):
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643021, Moscow
  - Investigational Site Number 643022, Novosibirsk
  - Investigational Site Number 643008, Saint Petersburg
  - Investigational Site Number 643010, Samara
- Investigational Site Number 703001, Košice, Slovakia
- South Korea (2):
  - Investigational Site Number 410017, Daejeon
  - Investigational Site Number 410016, Seoul
- Spain (9):
  - Investigational Site Number 724009, A Coruña
  - Investigational Site Number 724016, Barakaldo
  - Investigational Site Number 724015, Barcelona
  - Investigational Site Number 724014, Cadiz
  - Investigational Site Number 724001, Málaga
  - Investigational Site Number 724011, Sabadell
  - Investigational Site Number 724017, Santiago de Compostela
  - Investigational Site Number 724013, Santiago de Compostela
  - Investigational Site Number 724007, Seville
- Taiwan (3):
  - Investigational Site Number 158005, Kaohsiung City
  - Investigational Site Number 158006, Taipei
  - Investigational Site Number 158002, Taoyuan
- Turkey (Türkiye) (3):
  - Investigational Site Number 792007, Edirne
  - Investigational Site Number 792008, Gaziantep
  - Investigational Site Number 792009, Samsun
- Ukraine (5):
  - Investigational Site Number 804013, Kharkiv
  - Investigational Site Number 804014, Kyiv
  - Investigational Site Number 804027, Kyiv
  - Investigational Site Number 804011, Vinnytsia
  - Investigational Site Number 804009, Zaporizhzhya

REFERENCES:
- [Result] Fleischmann R, van Adelsberg J, Lin Y, Castelar-Pinheiro GD, Brzezicki J, Hrycaj P, Graham NM, van Hoogstraten H, Bauer D, Burmester GR. Sarilumab and Nonbiologic Disease-Modifying Antirheumatic Drugs in Patients With Active Rheumatoid Arthritis and Inadequate Response or Intolerance to Tumor Necrosis Factor Inhibitors. Arthritis Rheumatol. 2017 Feb;69(2):277-290. doi: 10.1002/art.39944. PMID 27860410
- [Derived] Choy E, Bykerk V, Lee YC, van Hoogstraten H, Ford K, Praestgaard A, Perrot S, Pope J, Sebba A. Disproportionate articular pain is a frequent phenomenon in rheumatoid arthritis and responds to treatment with sarilumab. Rheumatology (Oxford). 2023 Jul 5;62(7):2386-2393. doi: 10.1093/rheumatology/keac659. PMID 36413080
- [Derived] Rubbert-Roth A, Furst DE, Fiore S, Praestgaard A, Bykerk V, Bingham CO, Charles-Schoeman C, Burmester G. Association between low hemoglobin, clinical measures, and patient-reported outcomes in patients with rheumatoid arthritis: results from post hoc analyses of three phase III trials of sarilumab. Arthritis Res Ther. 2022 Aug 25;24(1):207. doi: 10.1186/s13075-022-02891-x. PMID 36008838
- [Derived] Rehberg M, Giegerich C, Praestgaard A, van Hoogstraten H, Iglesias-Rodriguez M, Curtis JR, Gottenberg JE, Schwarting A, Castaneda S, Rubbert-Roth A, Choy EHS; MOBILITY, MONARCH, TARGET, and ASCERTAIN investigators. Identification of a Rule to Predict Response to Sarilumab in Patients with Rheumatoid Arthritis Using Machine Learning and Clinical Trial Data. Rheumatol Ther. 2021 Dec;8(4):1661-1675. doi: 10.1007/s40744-021-00361-5. Epub 2021 Sep 14. PMID 34519964
- [Derived] Fleischmann R, Genovese MC, Maslova K, Leher H, Praestgaard A, Burmester GR. Long-term safety and efficacy of sarilumab over 5 years in patients with rheumatoid arthritis refractory to TNF inhibitors. Rheumatology (Oxford). 2021 Nov 3;60(11):4991-5001. doi: 10.1093/rheumatology/keab355. PMID 33871596
- [Derived] Genovese MC, Burmester GR, Hagino O, Thangavelu K, Iglesias-Rodriguez M, John GS, Gonzalez-Gay MA, Mandrup-Poulsen T, Fleischmann R. Interleukin-6 receptor blockade or TNFalpha inhibition for reducing glycaemia in patients with RA and diabetes: post hoc analyses of three randomised, controlled trials. Arthritis Res Ther. 2020 Sep 9;22(1):206. doi: 10.1186/s13075-020-02229-5. PMID 32907617
- [Derived] Genovese MC, Fleischmann R, Kivitz A, Lee EB, van Hoogstraten H, Kimura T, St John G, Mangan EK, Burmester GR. Efficacy and safety of sarilumab in combination with csDMARDs or as monotherapy in subpopulations of patients with moderately to severely active rheumatoid arthritis in three phase III randomized, controlled studies. Arthritis Res Ther. 2020 Jun 10;22(1):139. doi: 10.1186/s13075-020-02194-z. PMID 32522251
- [Derived] Gossec L, Strand V, Proudfoot C, Chen CI, Guillonneau S, Kimura T, van Hoogstraten H, Mangan E, Reaney M. Effects of Sarilumab on Rheumatoid Arthritis as Reported by Patients Using the Rheumatoid Arthritis Impact of Disease Scale. J Rheumatol. 2019 Oct;46(10):1259-1267. doi: 10.3899/jrheum.180904. Epub 2019 Mar 15. PMID 30877216
- [Derived] Gabay C, Msihid J, Zilberstein M, Paccard C, Lin Y, Graham NMH, Boyapati A. Identification of sarilumab pharmacodynamic and predictive markers in patients with inadequate response to TNF inhibition: a biomarker substudy of the phase 3 TARGET study. RMD Open. 2018 Mar 14;4(1):e000607. doi: 10.1136/rmdopen-2017-000607. eCollection 2018. PMID 29556418
- [Derived] Strand V, Reaney M, Chen CI, Proudfoot CW, Guillonneau S, Bauer D, Mangan E, Graham NM, van Hoogstraten H, Lin Y, Pacheco-Tena C, Fleischmann R. Sarilumab improves patient-reported outcomes in rheumatoid arthritis patients with inadequate response/intolerance to tumour necrosis factor inhibitors. RMD Open. 2017 Mar 7;3(1):e000416. doi: 10.1136/rmdopen-2016-000416. eCollection 2017. PMID 28326189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 240 centers in 27 countries. A total of 1224 participants were screened between 29 October 2012 and 7 August 2014, of whom 546 participants were randomized and 678 were screen failures. Screen failures were mainly due to failure to meet inclusion criteria.
Pre-assignment Details: Participants were randomized 1:1:1 (placebo q2w : sarilumab 150 mg q2w : sarilumab 200 mg q2w) via a centralized randomization system using an interactive voice response system stratified by region and number of previous anti- tumor necrosis factor (TNF) therapy (1 versus >1).
Groups:
- Placebo q2w: Placebo matched to sarilumab subcutaneous (SC) injection once every 2 weeks (q2w) was added to one or a combination of the nonbiologic disease modifying antirheumatic drug (DMARD) for 24 weeks.
- Sarilumab 150 mg q2w: Sarilumab 150 mg SC injection q2w was added to one or a combination of the nonbiologic DMARD for 24 weeks.
- Sarilumab 200 mg q2w: Sarilumab 200 mg SC injection q2w was added to one or a combination of the nonbiologic DMARD for 24 weeks.
Period: Overall Study
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Started | 181 | 181 | 184
Completed | 101 | 125 | 133
Not Completed | 80 | 56 | 51
Not completed — Rescued and entered in long term safety | 63 | 25 | 26
Not completed — Adverse Event | 9 | 18 | 17
Not completed — Lack of Efficacy | 5 | 4 | 2
Not completed — Poor compliance to protocol | 1 | 2 | 1
Not completed — Other, not related to safety or efficacy | 2 | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo q2w: Placebo matched to sarilumab SC injection q2w was added to one or a combination of the nonbiologic DMARD for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w | Total
Number analyzed (Participants) | 181 | 181 | 184 | 546
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (12.4) | 54.0 (11.7) | 52.9 (12.9) | 52.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 154 | 142 | 151 | 447
  Male | 27 | 39 | 33 | 99

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved at Least 20% Improvement in the American College of Rheumatology (ACR20) Criteria at Week 24
Description: ACR responses are assessed with a composite rating scale of the American College of Rheumatology that includes 7 variables: tender joint count (TJC); swollen joint count (SJC); levels of an acute phase reactant (C-reactive Protein levels [CRP]); participant's assessment of pain; participant's global assessment of disease activity; physician's global assessment of disease activity; participant's assessment of physical function by (health assessment questionnaire disability index [HAQ-DI]). ACR20 is defined as achieving at least 20% improvement in both TJC and SJC, and at least 20% improvement in at least 3 of the 5 other assessments of the ACR.
Time Frame: Week 24
Population: Intent-to-treat (ITT) population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
percentage of participants | 33.7 | 55.8 | 60.9
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; A hierarchical testing procedure was used to control type I error rate at 0.05 and handle multiple endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Threshold for significance at 0.025 level; Odds Ratio (OR) = 2.711, 95% CI 2-sided [1.730 to 4.247] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Threshold for significance at 0.025 level; Odds Ratio (OR) = 3.284, 95% CI 2-sided [2.108 to 5.115] — Sarilumab 200 mg q2w vs Placebo q2w

2. Primary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 12
Description: Physical function was assessed by HAQ-DI. It consisted of at least 2 questions per category, participant reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week rated on a 4-point scale where 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of category scores and divided by the number of categories answered, ranging from 0 to 3, where 0 = no disability and 3 = unable to do, high-dependency disability. Least-squares (LS) means and standard errors (SE) at Week 12 were obtained from a mixed-effect model with repeated measures (MMRM) with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline HAQ-DI as a covariate.
Time Frame: Baseline, Week 12
Population: ITT population. Number of participants analyzed = number of participants with HAQ-DI assessment at both baseline and Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 170 | 165 | 171
units on a scale | -0.26 (0.043) | -0.46 (0.044) | -0.47 (0.043)
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = -0.202, 95% CI 2-sided [-0.318 to -0.086] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = -0.210, 95% CI 2-sided [-0.325 to -0.095] — Sarilumab 200 mg q2w vs Placebo q2w

3. Secondary Outcome: Change From Baseline in Disease Activity Score for 28 Joints -C-Reactive Protein (DAS28--CRP) Score at Week 24
Description: DAS28 is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); General health (GH) assessment by the participant assessed from the ACR rheumatoid arthritis (RA) core set questionnaire (participant global assessment) in 100 mm visual analog scale (VAS). Marker of inflammation assessed by the high sensitivity C-reactive protein (hs-CRP) in mg/L. The DAS28 score provides a number indicating the current disease activity of the RA. DAS28 total score ranges from 2-10. A DAS28 score above 5.1 means high disease activity, whereas a DAS28 score below 3.2 indicates low disease activity and a DAS28 score below 2.6 means disease remission. LS means and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline DAS28-CRP score as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = number of participants with DAS28--CRP Score assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 99 | 126 | 136
units on a scale | -1.38 (0.119) | -2.35 (0.111) | -2.82 (0.108)
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = -0.971, 95% CI 2-sided [-1.283 to -0.658] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = -1.444, 95% CI 2-sided [-1.752 to -1.135] — Sarilumab 200 mg q2w vs Placebo q2w

4. Secondary Outcome: Percentage of Participants Achieving ACR50 Criteria at Week 24
Description: ACR responses are assessed with a composite rating scale that includes 7 variables: TJC; SJC; levels of an acute phase reactant (CRP level); participant's assessment of pain; participant's global assessment of disease activity; physician's global assessment of disease activity; participant's assessment of physical function by HAQ--DI. ACR50 is defined as achieving at least 50% improvement in both TJC and SJC, and at least 50% improvement in at least 3 of the 5 other assessments of the ACR.
Time Frame: Week 24
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
Percentage of participants | 18.2 | 37.0 | 40.8
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Threshold for significance at 0.025 level; Odds Ratio (OR) = 2.958, 95% CI 2-sided [1.764 to 4.959] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Threshold for significance was 0.025 level; Odds Ratio (OR) = 3.374, 95% CI 2-sided [2.045 to 5.566] — Sarilumab 200 mg q2w vs Placebo q2w

5. Secondary Outcome: Percentage of Participants Achieving ACR70 Criteria at Week 24
Description: ACR responses are assessed with a composite rating scale of the American College of Rheumatology that includes 7 variables: TJC; SJC; levels of an acute phase reactant (CRP level); participant's assessment of pain; participant's global assessment of disease activity; physician's global assessment of disease activity; participant's assessment of physical function by HAQ--DI. ACR70 is defined as achieving at least 70% improvement in both TJC and SJC, and at least 70% improvement in at least 3 of the 5 other assessments of the ACR.
Time Frame: Week 24
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
Percentage of participants | 7.2 | 19.9 | 16.3
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0002, Mantel Haenszel — Threshold for significance at 0.025 level; Odds Ratio (OR) = 3.607, 95% CI 2-sided [1.774 to 7.332] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0056, Mantel Haenszel — Threshold for significance at 0.025 level; Odds Ratio (OR) = 2.653, 95% CI 2-sided [1.308 to 5.383] — Sarilumab 200 mg q2w vs Placebo q2w

6. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Score (DAS28-CRP) <2.6 at Week 24
Description: DAS28 is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); GH by the participant assessed from the ACR rheumatoid arthritis core set questionnaire (participant global assessment) in 100 mm VAS; marker of inflammation assessed by hs-CRP in mg/L. The DAS28 provides a number indicating the current activity of the RA. DAS28 total score ranges from 2-10. A DAS28 score above 5.1 means high disease activity, whereas a DAS28 score below 3.2 indicates low disease activity and a DAS28 score below 2.6 means disease remission.
Time Frame: Week 24
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
Percentage of participants | 7.2 | 24.9 | 28.8
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Threshold for significance at 0.025 level; Odds Ratio (OR) = 4.622, 95% CI 2-sided [2.339 to 9.132] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Threshold for significance at 0.025 level; Odds Ratio (OR) = 5.801, 95% CI 2-sided [2.948 to 11.413] — Sarilumab 200 mg q2w vs Placebo q2w

7. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 24
Description: CDAI is a composite index constructed to measure clinical remission in RA that does not include a laboratory test, and is a numerical summation of 4 components: TJC (28 joints), SJC (28 joints), Participant's Global Assessment of Disease Activity VAS (in cm), and Physician's Global Assessment of Disease VAS (in cm). Total scores ranges from 0 to 76 with a negative change in CDAI score indicating an improvement in disease activity and a positive change in score indicating a worsening of disease activity. LS means and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline CDAI as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed=number of participants with CDAI assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 100 | 127 | 136
units on a scale | -16.35 (1.195) | -23.65 (1.136) | -26.08 (1.109)
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = -7.306, 95% CI 2-sided [-10.444 to -4.167] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = -9.727, 95% CI 2-sided [-12.833 to -6.622] — Sarilumab 200 mg q2w vs Placebo q2w

8. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24
Description: Physical function was assessed by HAQ-DI. It consisted of at least 2 questions per category, participant reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week rated on a 4-point scale where 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of category scores and divided by the number of categories answered, ranging from 0 to 3, where 0 = no disability and 3 = unable to do, high-dependency disability. LS means and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline HAQ-DI as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = number of participants with HAQ-DI assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 101 | 127 | 136
units on a scale | -0.34 (0.051) | -0.52 (0.049) | -0.58 (0.048)
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0078, Mixed Models Analysis — Threshold for significance was 0.025 level; LS Mean Difference = -0.183, 95% CI 2-sided [-0.318 to -0.048] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Threshold for significance was 0.025 level; LS Mean Difference = -0.242, 95% CI 2-sided [-0.376 to -0.109] — Sarilumab 200 mg q2w vs Placebo q2w

9. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Physical Component Summary Scores (PCS) at Week 24
Description: SF-36 is a generic 36-item questionnaire measuring health-related quality of life (HRQL) covering 2 summary measures: PCS and mental component summary (MCS). The SF-36 consists of 8 subscales. The PCS had 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception. The MCS had 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; 0= worst HRQL, 100=best HRQL. Higher scores indicate better health and well-being. LS mean and SE at Week 24 by MMRM with treatment,region,number of previous anti TNFs,visit,and treatment-by-visit interaction as fixed effects and baseline SF-36 (PCS) as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with SF-36 PCS assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 99 | 123 | 134
units on a scale | 4.40 (0.692) | 7.65 (0.653) | 8.48 (0.630)
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = 3.250, 95% CI 2-sided [1.450 to 5.049] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = 4.075, 95% CI 2-sided [2.305 to 5.846] — Sarilumab 200 mg q2w vs Placebo q2w

10. Secondary Outcome: Change From Baseline in SF-36 MCS at Week 24
Description: SF-36 is a generic 36-item questionnaire measuring HRQL covering 2 summary measures: PCS and MCS. The SF-36 consists of 8 subscales. The PCS is represented by 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; 0= worst HRQL, 100=best HRQL. Higher scores indicate better health and well-being. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline SF-36 MCS as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed=participants with SF-36 MCS assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 99 | 123 | 134
units on a scale | 4.74 (0.902) | 6.26 (0.848) | 6.76 (0.817)
Statistical Analysis 1: Comparison: Placebo q2w vs Sarilumab 150 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.2026, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = 1.515, 95% CI 2-sided [-0.818 to 3.848] — Sarilumab 150 mg q2w vs Placebo q2w
Statistical Analysis 2: Comparison: Placebo q2w vs Sarilumab 200 mg q2w; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0854, Mixed Models Analysis — Threshold for significance at 0.025 level; LS Mean Difference = 2.013, 95% CI 2-sided [-0.282 to 4.309] — Sarilumab 200 mg q2w vs Placebo q2w

11. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-fatigue) Score at Week 24
Description: The FACIT-Fatigue is a 13-item questionnaire assessing fatigue where participants scored each item on a 5-point scale (0-4): 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much. A total score ranging from 0 to 52. A higher score corresponded to a lower level of fatigue. A positive change from baseline score indicates an improvement. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline FACIT-fatigue as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of Participants analyzed = number of participants with FACIT-fatigue score assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 98 | 126 | 136
units on a scale | 6.82 (0.863) | 9.86 (0.802) | 10.06 (0.778)

12. Secondary Outcome: Change From Baseline in Morning Stiffness VAS at Week 24
Description: RA is associated with stiffness of joints, especially in the morning after prolonged stationery state. The degree of stiffness can be an indicator of disease severity. The severity of morning stiffness was assessed on a VAS scale from 0 mm (no problem) to 100 mm (major problem). LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline Morning Stiffness as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = number of participants with morning stiffness VAS assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 101 | 127 | 136
mm | -21.66 (2.390) | -32.30 (2.213) | -33.79 (2.148)

13. Secondary Outcome: Change From Baseline in Work Productivity Survey - Rheumatoid Arthritis (WPS-RA) at Week 24: Work Days Missed Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of work days missed in the last month by the participant was reported. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed=participants with WPS-RA individual items assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 32 | 43 | 45
Days | -2.01 (0.458) | -2.87 (0.438) | -3.19 (0.447)

14. Secondary Outcome: Change From Baseline in WPS-RA at Week 24: Days With Work Productivity Reduced by ≥ 50% Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of work days with reduced productivity by ≥ 50% in the last month by the participant was reported. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = participants with WPS-RA individual items assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 32 | 43 | 45
Days | -3.64 (0.589) | -4.26 (0.521) | -4.34 (0.535)

15. Secondary Outcome: Change From Baseline in WPS-RA at Week 24: RA Interference With Work Productivity
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Interference in the last month with work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference). LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 24
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 32 | 42 | 45
units on a scale | -1.632 (0.4186) | -2.422 (0.3719) | -2.727 (0.3700)

16. Secondary Outcome: Change From Baseline in WPS-RA at Week 24: House Work Days Missed Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with no household work in the last month by the participant was reported. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 24
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 101 | 126 | 133
Days | -3.50 (0.590) | -6.13 (0.551) | -6.18 (0.537)

17. Secondary Outcome: Change From Baseline in WPS-RA at Week 24: Days With Household Work Productivity Reduced by ≥ 50% Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with reduced household work productivity by ≥ 50% in the last month by the participant was reported. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 24
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 101 | 125 | 133
Days | -3.36 (0.632) | -4.60 (0.591) | -4.88 (0.574)

18. Secondary Outcome: Change From Baseline in WPS-RA at Week 24: Days With Family/Social/Leisure Activities Missed Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days missed of family/social/leisure activities in the last month by the participant was reported. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 24
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 101 | 127 | 133
Days | -1.97 (0.479) | -3.51 (0.446) | -4.12 (0.435)

19. Secondary Outcome: Change From Baseline in WPS-RA at Week 24: Days With Outside Help Hired Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with outside help hired in the last month by the participant was reported. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 24
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 101 | 126 | 133
Days | -1.60 (0.567) | -3.87 (0.536) | -3.86 (0.523)

20. Secondary Outcome: Change From Baseline in WPS-RA at Week 24: RA Interference With Household Work Productivity
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). The RA interference in the last month with household work productivity was measured on a scale that ranges from 0 (no interference) to 10 (complete interference). LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 24
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 100 | 126 | 132
units on a scale | -1.970 (0.2438) | -3.096 (0.2238) | -3.269 (0.2186)

21. Secondary Outcome: Change From Baseline in Rheumatoid Arthritis Impact of Disease (RAID) Scores at Week 24
Description: RAID is a composite measure of the impact of RA on participants that takes into account 7 domains: pain, functional disability, fatigue, physical and emotional well being, quality of sleep, and coping. The RAID is calculated based on 7 numerical rating scales (NRS) questions. Range of the final RAID value is 0-10 where 0= not affected, very good and 10 = most affected weighted and calculated with a total score range of 0 (not affected, very good) to 10 (most affected). A higher RAID value indicate worse status and lower indicate not affected. LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline RAID as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = number of participants with RAID score assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 99 | 126 | 136
units on a scale | -1.80 (0.203) | -2.55 (0.189) | -2.80 (0.183)

22. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimension 3 Level (EQ-5D-3L) VAS Scores at Week 24
Description: The EQ-5D-3L is a standardized, generic measure of health outcome. It was designed for self-completion by participants. It was specifically included to address concerns regarding the health economic impact of RA. The EQ-5D-3L comprises 5 questions on mobility, self-care, pain, usual activities, and psychological status with 3 possible answers for each item (1=no problem, 2=moderate problems, 3=severe problems) and a vertical VAS that allows the participants to indicate their health state today that can range from 0 (worst imaginable) to 100 (best imaginable). LS mean and SE at Week 24 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline EQ-5D-3L Scores as a covariate.
Time Frame: Baseline, Week 24
Population: ITT population. Number of participants analyzed = number of participants with EQ-5D-3L score assessment at both baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 96 | 126 | 133
units on a scale | 14.85 (2.098) | 20.06 (1.891) | 18.40 (1.842)

23. Secondary Outcome: Percentage of Participants Achieving ACR20, ACR50 and ACR70 Criteria at Week 12
Description: ACR responses are assessed with a composite rating scale of the American College of Rheumatology that includes 7 variables: TJC; SJC; levels of an acute phase reactant (CRP level); participant's assessment of pain; participant's global assessment of disease activity; physician's global assessment of disease activity; participant's assessment of physical function by HAQ--DI. ACR20 is defined as achieving at least 20% improvement in both TJC and SJC, and at least 20% improvement in at least 3 of the 5 other assessments of the ACR. ACR50 is defined as achieving at least 50% improvement in both TJC and SJC, and at least 50% improvement in at least 3 of the 5 other assessments of the ACR. ACR70 is defined as achieving at least 70% improvement in both TJC and SJC, and at least 70% improvement in at least 3 of the 5 other assessments of the ACR.
Time Frame: Week 12
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
Percentage of participants
  ACR20 | 37.6 | 54.1 | 62.5
  ACR50 | 13.3 | 30.4 | 33.2
  ACR70 | 2.2 | 13.8 | 14.7

24. Secondary Outcome: Change From Baseline in DAS28-CRP at Week 12
Description: DAS28 is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); GH by the participant assessed from the ACR rheumatoid arthritis core set questionnaire (participant global assessment) in 100 mm VAS; marker of inflammation assessed by hs-CRP in mg/L. The DAS28 provides a number indicating the current activity of the RA. DAS28 total score ranges from 2-10. A DAS28 score above 5.1 means high disease activity, whereas a DAS28 score below 3.2 indicates low disease activity and a DAS28 score below 2.6 means disease remission. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline DAS score as a covariate.
Time Frame: Baseline, Week 12
Population: ITT population. Number of participants analyzed = number of participants with DAS28-CRP- Score assessment at both baseline and Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 168 | 163 | 169
units on a scale | -0.97 (0.104) | -2.13 (0.105) | -2.45 (0.103)

25. Secondary Outcome: Percentage of Participants Achieving Clinical Remission Score (DAS28--CRP <2.6) at Week 12
Description: DAS28 is a composite score that includes 4 variables: TJC (based on 28 joints); SJC (based on 28 joints); GH by the participant assessed from the ACR RA core set questionnaire (participant global assessment) in 100 mm VAS; marker of inflammation assessed by hs-CRP in mg/L. The DAS28 provides a number indicating the current activity of the RA. DAS28 total score ranges from 2-10. A DAS28 score above 5.1 means high disease activity, whereas a DAS28 score below 3.2 indicates low disease activity and a DAS28 score below 2.6 means disease remission.
Time Frame: Week 12
Population: ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
Percentage of participants | 3.9 | 17.1 | 17.9

26. Secondary Outcome: Change From Baseline in SF-36 at Week 12
Description: SF-36 is a generic 36-item questionnaire measuring HRQL covering 2 summary measures: PCS and MCS. The SF-36 consists of 8 subscales. The PCS is represented by 4 subscales: physical function, role limitations due to physical problems, pain, and general health perception. The MCS is represented by 4 subscales: vitality, social function, role limitations due to emotional problems, and mental health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; 0= worst HRQL, 100=best HRQL. Higher scores indicate better health and well-being. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline SF-36 as a covariate.
Time Frame: Baseline, Week 12
Population: ITT population. Number of participants analyzed=participants with SF-36 assessment at both baseline and Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 169 | 160 | 165
units on a scale
  Physical Component Summary Score at Week 12 | 3.74 (0.582) | 6.93 (0.596) | 6.84 (0.584)
  Mental Component Summary Score at Week 12 | 3.50 (0.738) | 5.14 (0.758) | 6.47 (0.741)

27. Secondary Outcome: Change From Baseline in WPS-RA at Week 12: Work Days Missed Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of work days missed in the last month by the participant was reported. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 12
Population: ITT population. Number of participants analyzed=participants with WPS-RA individual items assessment at both baseline and Week 12.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 54 | 54 | 56
Days | -1.20 (0.581) | -1.97 (0.571) | -2.98 (0.585)

28. Secondary Outcome: Change From Baseline in WPS-RA at Week 12: Days With Work Productivity Reduced by ≥ 50% Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of work days with reduced productivity by ≥ 50% in the last month by the participant was reported. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 12
Population: ITT population. Number of participants analyzed = participants with WPS-RA individual items assessment at both baseline and Week 12.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 54 | 54 | 56
Days | -1.69 (0.784) | -4.24 (0.773) | -3.20 (0.785)

29. Secondary Outcome: Change From Baseline in WPS-RA at Week 12: RA Interference With Work Productivity
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Interference in the last month with work productivity was measured on a scale that ranges from 0 (no interference) to 10 (complete interference). LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 12
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 53 | 54 | 56
units on a scale | -1.043 (0.3803) | -1.924 (0.3742) | -1.873 (0.3764)

30. Secondary Outcome: Change From Baseline in WPS-RA at Week 12: House Work Days Missed Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with no household work in the last month by the participant was reported. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 12
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 170 | 164 | 169
Days | -2.10 (0.551) | -5.52 (0.563) | -5.54 (0.553)

31. Secondary Outcome: Change From Baseline in WPS-RA at Week 12: Days With Household Work Productivity Reduced by ≥ 50% Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with reduced household work productivity by ≥ 50% in the last month by the participant was reported. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 12
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 169 | 163 | 169
Days | -2.60 (0.576) | -3.97 (0.587) | -3.98 (0.575)

32. Secondary Outcome: Change From Baseline in WPS-RA at Week 12: Days With Family/Social/Leisure Activities Missed Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days missed of family/social/leisure activities in the last month by the participant was reported. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 12
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 170 | 164 | 169
Days | -2.23 (0.433) | -2.53 (0.442) | -3.26 (0.434)

33. Secondary Outcome: Change From Baseline in WPS-RA at Week 12: Days With Outside Help Hired Due to RA
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). Number of days with outside help hired in the last month by the participant was reported. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 12
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 170 | 164 | 169
Days | -0.77 (0.558) | -3.07 (0.570) | -2.94 (0.560)

34. Secondary Outcome: Change From Baseline in WPS-RA at Week 12: RA Interference With Household Work Productivity
Description: The WPS-RA is a validated questionnaire that evaluates productivity limitations within work and within home associated with RA over the previous month. The questionnaire was interviewer-administered and was based on participant self-report. It contains 9 questions addressing employment status (1 item), productivity at work (3 items), and within and outside the home (5 items). The RA interference in the last month with household work productivity was measured on a scale that ranges from 0 (no interference) to 10 (complete interference). LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline WPS-RA as a covariate.
Time Frame: Baseline, Week 12
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 169 | 164 | 167
units on a scale | -1.210 (0.2428) | -2.772 (0.2474) | -2.404 (0.2443)

35. Secondary Outcome: Change From Baseline in the FACIT-fatigue at Week 12
Description: The FACIT-Fatigue is a 13-item questionnaire assessing fatigue where participants scored each item on a 5-point scale (0-4): 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much. A total score ranging from 0 to 52. A higher score corresponded to a lower level of fatigue. A positive change from baseline score indicates an improvement. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline FACIT-fatigue as a covariate.
Time Frame: Baseline, Week 12
Population: ITT population. Number of Participants analyzed = number of participants with FACIT-fatigue score assessment at both baseline and Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 169 | 165 | 172
units on a scale | 5.56 (0.721) | 8.02 (0.729) | 9.45 (0.714)

36. Secondary Outcome: Change From Baseline in EQ-5D-3L VAS Scores at Week 12
Description: The EQ-5D-3L is a standardized, generic measure of health outcome. EQ-5D was designed for self-completion by participants. The EQ-5D was specifically included to address concerns regarding the health economic impact of RA. The EQ-5D-3L comprises 5 questions on mobility, self-care, pain, usual activities, and psychological status with 3 possible answers for each item (1=no problem, 2=moderate problems, 3=severe problems) and a vertical VAS that allows the participants to indicate their health state today that can range from 0 (worst imaginable) to 100 (best imaginable). LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline EQ-5D-3L scores as a covariate.
Time Frame: Baseline, Week 12
Population: ITT population. Number of participants analyzed = number of participants with EQ-5D-3L score assessment at both baseline and Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 167 | 163 | 171
units on a scale | 8.39 (1.699) | 17.16 (1.720) | 15.23 (1.680)

37. Secondary Outcome: Change From Baseline in RAID Scores at Week 12
Description: RAID score is a composite measure of the impact of RA on participants that takes into account 7 domains: pain, functional disability, fatigue, physical and emotional well being, quality of sleep, and coping. The RAID is calculated based on 7 NRS questions. Range of the final RAID value is 0-10 where 0= not affected, very good and 10 = most affected weighted and calculated with a total score range of 0 (not affected, very good) to 10 (most affected). A higher RAID value indicates worse status and lower indicates not affected. LS mean and SE at Week 12 were obtained from a MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline RAID scores as a covariate.
Time Frame: Baseline, Week 12
Population: ITT population. Number of participants analyzed = number of participants with RAID score assessment at both baseline and Week 12.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 167 | 162 | 171
units on a scale | -1.34 (0.163) | -2.27 (0.165) | -2.47 (0.161)

38. Secondary Outcome: Change From Baseline in Individual ACR Components - TJC and SJC at Week 12 and Week 24
Description: ACR components were: TJC, SJC, physician global VAS, participant global VAS, pain VAS,HAQ-DI & CRP. 68 joints were assessed for tenderness (TJC scoring 0-68) and 66 joints for swelling (SJC scoring 0-66). The 66 SJC evaluated the following joints: temporomandibular, sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeal, interphalangeal of thumb, distal interphalangeal, proximal interphalangeal, knee, ankle mortise, ankle tarsus, metatarsophalangeal, interphalangeal of great toe, and proximal/distal interphalangeal of the toes. The TJC examined hip joints, in addition to the joints assessed for SJC. Increase in number of tender joints/swollen joints indicated severity. LS mean and SE at Week 12 & 24 by MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline ACR components as a covariate.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Number analyzed = number of participants with TJC and SJC assessments at both baseline and specified time points.
Measure: Least Squares Mean (Standard Error); unit: joints
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
joints
  TJC at week 12: number analyzed (Participants) | 172 | 165 | 172
  TJC at week 12 | -8.55 (0.959) | -13.74 (0.975) | -14.87 (0.954)
  SJC at week 12: number analyzed (Participants) | 172 | 165 | 172
  SJC at week 12 | -6.75 (0.687) | -10.54 (0.698) | -10.59 (0.684)
  TJC at week 24: number analyzed (Participants) | 101 | 127 | 137
  TJC at week 24 | -10.55 (1.060) | -14.44 (1.017) | -16.95 (0.992)
  SJC at week 24: number analyzed (Participants) | 101 | 127 | 137
  SJC at week 24 | -8.19 (0.721) | -11.56 (0.691) | -11.94 (0.674)

39. Secondary Outcome: Change From Baseline in Individual ACR Component - Physician Global VAS, Participant Global VAS and Pain VAS at Week 12 and Week 24
Description: ACR components were: TJC, SJC, physician global VAS, participant global VAS, pain VAS, HAQ-DI & CRP. Physician global VAS & participant global VAS was done by 100 mm non-anchored VAS, from no arthritis (0) activity to maximal arthritis (100) activity. Pain VAS by 100 mm VAS ranging from 0 "no pain" to 100 "worst pain". LS mean and SE at Week 12 & 24 by MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline ACR components as a covariate.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Number analyzed = number of participants with individual ACR components assessment at both baseline and specified time points.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
mm
  Physician global VAS at week 12: number analyzed (Participants) | 172 | 165 | 171
  Physician global VAS at week 12 | -22.74 (1.744) | -33.64 (1.775) | -35.44 (1.740)
  Participant global VAS at week 12: number analyzed (Participants) | 172 | 165 | 171
  Participant global VAS at week 12 | -13.75 (1.807) | -25.28 (1.836) | -27.38 (1.803)
  Pain VAS at week 12: number analyzed (Participants) | 171 | 166 | 171
  Pain VAS at week 12 | -15.13 (1.908) | -26.93 (1.933) | -30.56 (1.901)
  Physician global VAS at week 24: number analyzed (Participants) | 101 | 127 | 137
  Physician global VAS at week 24 | -28.55 (1.806) | -40.65 (1.695) | -43.22 (1.646)
  Participant global VAS at week 24: number analyzed (Participants) | 100 | 127 | 136
  Participant global VAS at week 24 | -19.76 (2.171) | -29.59 (2.046) | -31.28 (1.997)
  Pain VAS at week 24: number analyzed (Participants) | 98 | 127 | 135
  Pain VAS at week 24 | -21.27 (2.250) | -31.90 (2.086) | -33.65 (2.037)

40. Secondary Outcome: Change From Baseline in Individual ACR Component - CRP Level at Week 12 and Week 24
Description: ACR components were: TJC, SJC, physician global VAS, participant global VAS, pain VAS, HAQ-DI & CRP. An elevated CRP level was considered a non-specific "marker" for RA. A reduction level indicates improvement. LS mean and SE at Week 12 & 24 by MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline ACR components as a covariate.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Number analyzed = number of participants with CRP assessment at both baseline and specified time points.
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
mg/L
  CRP at week 12: number analyzed (Participants) | 168 | 165 | 170
  CRP at week 12 | -3.63 (1.436) | -15.08 (1.452) | -22.98 (1.432)
  CRP at week 24: number analyzed (Participants) | 100 | 126 | 137
  CRP at week 24 | -3.60 (1.556) | -15.24 (1.457) | -23.27 (1.421)

41. Secondary Outcome: Change From Baseline in Individual ACR Component - HAQ-DI at Week 12 and Week 24
Description: ACR components were: TJC, SJC, physician global VAS, participant global VAS, pain VAS,HAQ-DI & CRP. HAQ-DI consisted of at least 2 questions per category, participant reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week rated on a 4-point scale where 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of category scores and divided by the number of categories answered, ranging from 0 to 3, where 0 = no disability and 3 = unable to do, high-dependency disability. LS mean and SE at Week 12 & 24 by MMRM with treatment, region, number of previous anti-TNFs, visit, and treatment-by-visit interaction as fixed effects and baseline ACR components as a covariate.
Time Frame: Baseline, Week 12 and Week 24
Population: ITT population. Number analyzed = number of participants with HAQ-DI assessment at both baseline and specified time points.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 181 | 181 | 184
units on a scale
  HAQ-DI at week 12: number analyzed (Participants) | 170 | 165 | 171
  HAQ-DI at week 12 | -0.26 (0.043) | -0.46 (0.044) | -0.47 (0.043)
  HAQ-DI at week 24: number analyzed (Participants) | 101 | 127 | 136
  HAQ-DI at week 24 | -0.34 (0.051) | -0.52 (0.049) | -0.58 (0.048)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 30) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent AEs that is AEs that developed/worsened during the 'on treatment period' (time from the first dose injection of study drug to the end of follow-up period). Safety population included all participants from the randomized population who received at least 1 dose or part of a dose of study drug.
Arm/Group | Placebo q2w | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Serious Adverse Events (participants affected / at risk) | 6/181 | 6/181 | 10/184
Other Adverse Events (participants affected / at risk) | 26/181 | 60/181 | 57/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo q2w (N=181) | Sarilumab 150 mg q2w (N=181) | Sarilumab 200 mg q2w (N=184)
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 1
Endocarditis noninfective (Cardiac disorders) | 0 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Mixed liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo q2w (N=181) | Sarilumab 150 mg q2w (N=181) | Sarilumab 200 mg q2w (N=184)
Nasopharyngitis (Infections and infestations) | 9 | 11 | 7
Urinary tract infection (Infections and infestations) | 12 | 6 | 13
Neutropenia (Blood and lymphatic system disorders) | 2 | 23 | 22
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 11 | 5
Injection site erythema (General disorders) | 0 | 11 | 7
Alanine aminotransferase increased (Investigations) | 2 | 5 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.